CLINICAL TRIAL: NCT05792527
Title: The Use of L-carnitine in Modulating Pain and Inflammation in Rheumatoid Arthritis Patients
Brief Title: L-carnitine in Modulating Pain and Inflammation in Rheumatoid Arthritis
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Abdallah Abo-Elazm Shebl Eldisouky, principal investigator, Tanta University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: L-carnitine in RA
Record Dates: First submitted 2023-03-19; First posted 2023-03-31 (Actual); Last update posted 2023-03-31 (Actual); Status verified 2023-03

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Carnitine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (No Intervention): this group will include 23 patients which will receive the traditional therapy of RA for 3 months.
- L-carnitine group (Active Comparator): this group will include 23 patients which will receive 500mg L-carnitine two times daily after meal plus the traditional therapy of RA for 3 months.
  Interventions: Drug: L-carnitine

INTERVENTIONS:
Drug: L-carnitine — One 500 mg tablet twice daily after meals
  Arms: L-carnitine group

SUMMARY:
This study aims at evaluating the possible efficacy and safety of L-carnitine in rheumatoid arthritis via targeting Jak/STAT pathway and TGF-β1

ELIGIBILITY:
Inclusion Criteria:

* Patients with active rheumatoid arthritis (not in remission) according to American College of Rheumatology/European League Against Rheumatism (ACR/EULAR) 2010 criteria (9) i.e., 28 joints disease activity score (DAS-28) >2.6.
* Patients receive the conventional DMARDs
* Both sexes.
* Age range between 18 and 70 years old.

Exclusion Criteria:

* Patients with heart disease (congestive heart failure, arrhythmia, hypertension, ischemic heart diseases), diabetes, active infection, other illness except rheumatoid arthritis.
* Patients with renal and hepatic dysfunction.
* Patients receiving biological DMARDs.
* Patients receiving oral prednisolone greater than 15 mg/day.
* Patients with hypersensitivity to study medications.
* Patients using antioxidants.
* Pregnant and lactating females.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2023-03-05 (Actual); Primary Completion 2025-03-05 (Estimated); Study Completion 2026-03-05 (Estimated)

PRIMARY OUTCOMES:
The change in DAS-28-CRP score | 3 months
  Patients will undergo clinical assessment according to DAS-28-CRP score
The change in Multidimensional Health Assessment Questionnaire (MDHAQ) score | 3 months

SECONDARY OUTCOMES:
The change in serum level of C-reactive protein (CRP) | 3 months
  Blood samples will be collected at base line and after 3 months
The change in serum level of Signal transducer and activator of transcription 3(STAT 3). | 3 months
  Blood samples will be collected at base line and after 3 months
The change in serum level of Transforming growth factor β1(TGF-β1). | 3 months
  Blood samples will be collected at base line and after 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta university, Tanta, Gharbia Governorate, Egypt